CLINICAL TRIAL: NCT04799613
Title: Experimentally-induced Freezing of Gait in Parkinson's Disease by Modulating Step Length/Asymmetry and Cognitive/Visual Loading
Brief Title: Provocation of Freezing of Gait in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Alfonso Fasano, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 19-6049-B
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease; Freezing of Gait
Keywords: Parkinson; freezing; spilt-belt; Dual task; visual
MeSH Terms: conditions — Parkinson Disease | interventions — Walking Speed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Natural walking (No Intervention)
- fast walking (Experimental)
  Interventions: Other: walking speed
- normal walking passing through narrow pathway (Experimental)
  Interventions: Other: visual loading
- fast walking passing through narrow pathway (Experimental)
  Interventions: Other: walking speed; Other: visual loading
- Natural walking with dual task (Experimental)
  Interventions: Other: dual task
- fast walking with dual task (Experimental)
  Interventions: Other: walking speed; Other: dual task
- Natural walking passing through narrow pathway and during cognitive dual task (Experimental)
  Interventions: Other: visual loading; Other: dual task
- fast walking passing through narrow pathway and during cognitive dual task (Experimental)
  Interventions: Other: walking speed; Other: visual loading; Other: dual task
- Natural walking reducing the best side (Experimental)
  Interventions: Other: best side reduction
- fast walking reducing the best side (Experimental)
  Interventions: Other: walking speed; Other: best side reduction
- Natural walking reducing the best side passing through narrow pathway (Experimental)
  Interventions: Other: visual loading; Other: best side reduction
- fast walking reducing the best side passing through narrow pathway (Experimental)
  Interventions: Other: walking speed; Other: visual loading; Other: best side reduction
- Natural walking reducing the best side with cognitive dual task (Experimental)
  Interventions: Other: dual task; Other: best side reduction
- fast walking reducing the best side with cognitive dual task (Experimental)
  Interventions: Other: walking speed; Other: dual task; Other: best side reduction
- Natural walking reducing the best side passing through narrow pathway and during cognitive dual task (Experimental)
  Interventions: Other: visual loading; Other: dual task; Other: best side reduction
- fast walking reducing the best side passing through narrow pathway and during cognitive dual task (Experimental)
  Interventions: Other: walking speed; Other: visual loading; Other: dual task; Other: best side reduction

INTERVENTIONS:
Other: walking speed — walking speed (normal speed vs. fast speed). fast speed was 25% faster than normal speed
  Arms: fast walking; fast walking passing through narrow pathway; fast walking passing through narrow pathway and during cognitive dual task; fast walking reducing the best side; fast walking reducing the best side passing through narrow pathway; fast walking reducing the best side passing through narrow pathway and during cognitive dual task; fast walking reducing the best side with cognitive dual task; fast walking with dual task
Other: visual loading — visual loading (walking through narrow pathway using VR)
  Arms: Natural walking passing through narrow pathway and during cognitive dual task; Natural walking reducing the best side passing through narrow pathway; Natural walking reducing the best side passing through narrow pathway and during cognitive dual task; fast walking passing through narrow pathway; fast walking passing through narrow pathway and during cognitive dual task; fast walking reducing the best side passing through narrow pathway; fast walking reducing the best side passing through narrow pathway and during cognitive dual task; normal walking passing through narrow pathway
Other: dual task — dual task (serial subtraction using VR)
  Arms: Natural walking passing through narrow pathway and during cognitive dual task; Natural walking reducing the best side passing through narrow pathway and during cognitive dual task; Natural walking reducing the best side with cognitive dual task; Natural walking with dual task; fast walking passing through narrow pathway and during cognitive dual task; fast walking reducing the best side passing through narrow pathway and during cognitive dual task; fast walking reducing the best side with cognitive dual task; fast walking with dual task
Other: best side reduction — best side reduction (split belt mode, the speed of best side was reduced by 25% compared to the other side)
  Arms: Natural walking reducing the best side; Natural walking reducing the best side passing through narrow pathway; Natural walking reducing the best side passing through narrow pathway and during cognitive dual task; Natural walking reducing the best side with cognitive dual task; fast walking reducing the best side; fast walking reducing the best side passing through narrow pathway; fast walking reducing the best side passing through narrow pathway and during cognitive dual task; fast walking reducing the best side with cognitive dual task

SUMMARY:
Sample Size N= 10 Parkinson's disease patients with self-reported freezing of gait and 10 without self-reported freezing of gait (in total, 20 Parkinson's disease patients)

Accrual Period Single visit for 2 hours

Study Design This is a cross-sectional study with an intervention to provoke freezing of gait using split-belt treadmill in Parkinson's disease patients with a randomized cross-over design.

After baseline evaluation (a), interventions to induce freezing of gait will be performed in a randomized order to avoid a practice/fatigue effect in the following conditions using combination of 4 interventions: walking speed (fast walking vs. natural walking), visual loading (passing through narrow pathway), cognitive loading (dual task), and asymmetry (best side reduction).

1. Natural and fast walking with self-paced mode to access gait parameters and decide the speed for evaluation (3 mins X2) remaining assessment will be randomized and performed on the treadmill:
2. Natural and fast walking passing through narrow pathway (2 mins X2)
3. Natural and fast walking with dual task (2 mins X2)
4. Natural and fast walking passing through narrow pathway and during cognitive dual task (2 mins X2)
5. Natural and fast walking reducing the best side (2 mins X2)
6. Natural and fast walking reducing the best side passing through narrow pathway (2 mins X2)
7. Natural and fast walking reducing the best side with cognitive dual task (2 mins X2)
8. Natural and fast walking reducing the best side passing through narrow pathway and during cognitive dual task (2 mins X2)

   * Conditions b-h will be carried out on a split-belt treadmill (Grail systems®, by Motek, Netherlands).
   * (b-i) freezing of gait episodes will be identified with synchronized videorecordings (screening done by two independent observers). Episodes identified by both observers will be confirmed and measured by comparing the relative height of metatarsal and heel markers of each foot, in keeping with a previous study evaluating freezing of gait episode on a treadmill.

Study Duration

1. (Baselines evaluation) Enrolment and assessment (Montreal cognitive assessment, Movement Disorders Society-unified Parkinson's disease rating scale part 2, 3 and 4, Activities-Specific Balance Confidence Scale, Parkinson's disease questionnaire-39, and New freezing of gait questionnaire)
2. (a) Formal gait analysis using split-belt treadmill (Grail systems®, by Motek, Netherlands) will be done for baseline assessment (normal walking) and to test patient's ability for fast walking (25% of the normal speed).
3. (b-h) Provocation of freezing of gait at split-belt treadmill (Grail systems®, by Motek, Netherlands) with natural and fast walking with/without additional loading or interventions on the asymmetry

Total time= 2 hours

Study Intervention Freezing of gait will be provoked based on the situations combined among 4 conditions; (1) interventions on asymmetry, (2) cognitive dual task, (3) visual loading - passing through narrow pathway, and (4) walking speed at a split-belt treadmill.

* Fast walking will be defined as walking 25% faster than the normal comfortable walking. Subjects who cannot reach this speed, will be asked to walk at their safest maximum speed.
* Passing narrow pathway will be done by walking in a "rope bridge" scene in virtual reality (VR).
* Dual cognitive task will be carried out with serial subtraction prompted on the screen in VR.
* Best side reduction will be defined as 25% slower speed on the best side based on the speed during the initial natural walking with tied configuration setting based on a previous study.3
* Condition b-h will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease
* Hoehn & Yahr Stage 1-3
* Ten with self-reported freezing of gait (score of 1 in part 1 of new freezing of gait questionnaire), and 10 without FOG..
* Sequence effect on feet (as score of at least 2 in the leg agility (item#3.8) of Movement Disorders Society-Unified Parkinson's disease rating scale part 3)
* Stable clinical response to medications or stimulation parameters for at least 1 months
* Able to walk on a motor-driven treadmill
* Ability to provide informed consent

Exclusion Criteria:

* Severe imbalance that limits ambulation (Hoehn &Yahr score above 4)
* Orthostatic hypotension
* Orthopedic conditions and other systemic disease affecting locomotion
* Shortness of breath and cardiac disease
* Psychiatric disorders needing medication
* Dementia
* Presence of other neurological disorder

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
number of freezing of gait | Within intervention (2mins for each situation)
  provoked freezing of gait during each situation

SECONDARY OUTCOMES:
Correlation with Montreal cognitive assessment, Movement Disorders Society-unified Parkinson's disease rating scale part 2 and 3, Activities-Specific Balance Confidence Scale, Parkinson's disease questionnaire-39, and New freezing of gait questionnaire | Within intervention (2mins for each situation)
  Correlation of detected number of freezing of gait with clinical scales
Comparison of number/duration of provoked freezing of gait among the situations between Parkinson's disease patients with and without freezing of gait | Within intervention (2mins for each situation)
  Comparison between two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nieuwboer A, Rochester L, Herman T, Vandenberghe W, Emil GE, Thomaes T, Giladi N. Reliability of the new freezing of gait questionnaire: agreement between patients with Parkinson's disease and their carers. Gait Posture. 2009 Nov;30(4):459-63. doi: 10.1016/j.gaitpost.2009.07.108. Epub 2009 Aug 5. PMID 19660949
- [Background] Fasano A, Herzog J, Seifert E, Stolze H, Falk D, Reese R, Volkmann J, Deuschl G. Modulation of gait coordination by subthalamic stimulation improves freezing of gait. Mov Disord. 2011 Apr;26(5):844-51. doi: 10.1002/mds.23583. Epub 2011 Mar 2. PMID 21370271
- [Background] Fasano A, Schlenstedt C, Herzog J, Plotnik M, Rose FEM, Volkmann J, Deuschl G. Split-belt locomotion in Parkinson's disease links asymmetry, dyscoordination and sequence effect. Gait Posture. 2016 Jul;48:6-12. doi: 10.1016/j.gaitpost.2016.04.020. Epub 2016 Apr 27. PMID 27477701
- [Background] Giladi N, Kao R, Fahn S. Freezing phenomenon in patients with parkinsonian syndromes. Mov Disord. 1997 May;12(3):302-5. doi: 10.1002/mds.870120307. PMID 9159723
- [Background] Giladi N, Treves TA, Simon ES, Shabtai H, Orlov Y, Kandinov B, Paleacu D, Korczyn AD. Freezing of gait in patients with advanced Parkinson's disease. J Neural Transm (Vienna). 2001;108(1):53-61. doi: 10.1007/s007020170096. PMID 11261746
- [Background] Chee R, Murphy A, Danoudis M, Georgiou-Karistianis N, Iansek R. Gait freezing in Parkinson's disease and the stride length sequence effect interaction. Brain. 2009 Aug;132(Pt 8):2151-60. doi: 10.1093/brain/awp053. Epub 2009 May 11. PMID 19433440
- [Background] Plotnik M, Giladi N, Balash Y, Peretz C, Hausdorff JM. Is freezing of gait in Parkinson's disease related to asymmetric motor function? Ann Neurol. 2005 May;57(5):656-63. doi: 10.1002/ana.20452. PMID 15852404
- [Background] Youn J, Okuma Y, Hwang M, Kim D, Cho JW. Falling Direction can Predict the Mechanism of Recurrent Falls in Advanced Parkinson's Disease. Sci Rep. 2017 Jun 20;7(1):3921. doi: 10.1038/s41598-017-04302-7. PMID 28634343
- [Background] Giladi N. Medical treatment of freezing of gait. Mov Disord. 2008;23 Suppl 2:S482-8. doi: 10.1002/mds.21914. PMID 18668620
- [Background] Sawada M, Wada-Isoe K, Hanajima R, Nakashima K. Clinical features of freezing of gait in Parkinson's disease patients. Brain Behav. 2019 Apr;9(4):e01244. doi: 10.1002/brb3.1244. Epub 2019 Mar 9. PMID 30851088
- [Background] Snijders AH, Weerdesteyn V, Hagen YJ, Duysens J, Giladi N, Bloem BR. Obstacle avoidance to elicit freezing of gait during treadmill walking. Mov Disord. 2010 Jan 15;25(1):57-63. doi: 10.1002/mds.22894. PMID 19938174
- [Background] Spildooren J, Vercruysse S, Desloovere K, Vandenberghe W, Kerckhofs E, Nieuwboer A. Freezing of gait in Parkinson's disease: the impact of dual-tasking and turning. Mov Disord. 2010 Nov 15;25(15):2563-70. doi: 10.1002/mds.23327. PMID 20632376
- [Background] Ginis P, Nackaerts E, Nieuwboer A, Heremans E. Cueing for people with Parkinson's disease with freezing of gait: A narrative review of the state-of-the-art and novel perspectives. Ann Phys Rehabil Med. 2018 Nov;61(6):407-413. doi: 10.1016/j.rehab.2017.08.002. Epub 2017 Sep 7. PMID 28890341
- [Background] Lu C, Amundsen Huffmaster SL, Tuite PJ, Vachon JM, MacKinnon CD. Effect of Cue Timing and Modality on Gait Initiation in Parkinson Disease With Freezing of Gait. Arch Phys Med Rehabil. 2017 Jul;98(7):1291-1299.e1. doi: 10.1016/j.apmr.2017.01.009. Epub 2017 Feb 4. PMID 28167093
- [Background] Nutt JG, Bloem BR, Giladi N, Hallett M, Horak FB, Nieuwboer A. Freezing of gait: moving forward on a mysterious clinical phenomenon. Lancet Neurol. 2011 Aug;10(8):734-44. doi: 10.1016/S1474-4422(11)70143-0. PMID 21777828
- [Background] Nonnekes J, Bloem BR. Biphasic Levodopa-Induced Freezing of Gait in Parkinson's Disease. J Parkinsons Dis. 2020;10(3):1245-1248. doi: 10.3233/JPD-201997. PMID 32417798
- [Background] Barbe MT, Amarell M, Snijders AH, Florin E, Quatuor EL, Schonau E, Fink GR, Bloem BR, Timmermann L. Gait and upper limb variability in Parkinson's disease patients with and without freezing of gait. J Neurol. 2014 Feb;261(2):330-42. doi: 10.1007/s00415-013-7199-1. Epub 2013 Dec 4. PMID 24305993
- [Background] Hausdorff JM, Schaafsma JD, Balash Y, Bartels AL, Gurevich T, Giladi N. Impaired regulation of stride variability in Parkinson's disease subjects with freezing of gait. Exp Brain Res. 2003 Mar;149(2):187-94. doi: 10.1007/s00221-002-1354-8. Epub 2003 Jan 22. PMID 12610686
- [Background] Nanhoe-Mahabier W, Snijders AH, Delval A, Weerdesteyn V, Duysens J, Overeem S, Bloem BR. Split-belt locomotion in Parkinson's disease with and without freezing of gait. Neuroscience. 2013 Apr 16;236:110-6. doi: 10.1016/j.neuroscience.2013.01.038. Epub 2013 Jan 29. PMID 23370318
- [Background] Ricciardi L, Ricciardi D, Lena F, Plotnik M, Petracca M, Barricella S, Bentivoglio AR, Modugno N, Bernabei R, Fasano A. Working on asymmetry in Parkinson's disease: randomized, controlled pilot study. Neurol Sci. 2015 Aug;36(8):1337-43. doi: 10.1007/s10072-015-2082-8. Epub 2015 Feb 13. PMID 25677846
- [Background] Seuthe J, D'Cruz N, Ginis P, Becktepe JS, Weisser B, Nieuwboer A, Schlenstedt C. The Effect of One Session Split-Belt Treadmill Training on Gait Adaptation in People With Parkinson's Disease and Freezing of Gait. Neurorehabil Neural Repair. 2020 Oct;34(10):954-963. doi: 10.1177/1545968320953144. Epub 2020 Sep 17. PMID 32940131
- [Background] D'Cruz N, Seuthe J, Ginis P, Hulzinga F, Schlenstedt C, Nieuwboer A. Short-Term Effects of Single-Session Split-Belt Treadmill Training on Dual-Task Performance in Parkinson's Disease and Healthy Elderly. Front Neurol. 2020 Sep 30;11:560084. doi: 10.3389/fneur.2020.560084. eCollection 2020. PMID 33101174
- [Background] Berardelli A, Rothwell JC, Thompson PD, Hallett M. Pathophysiology of bradykinesia in Parkinson's disease. Brain. 2001 Nov;124(Pt 11):2131-46. doi: 10.1093/brain/124.11.2131. PMID 11673316
- [Background] Bologna M, Guerra A, Paparella G, Giordo L, Alunni Fegatelli D, Vestri AR, Rothwell JC, Berardelli A. Neurophysiological correlates of bradykinesia in Parkinson's disease. Brain. 2018 Aug 1;141(8):2432-2444. doi: 10.1093/brain/awy155. PMID 29901693
- [Background] Iansek R, Huxham F, McGinley J. The sequence effect and gait festination in Parkinson disease: contributors to freezing of gait? Mov Disord. 2006 Sep;21(9):1419-24. doi: 10.1002/mds.20998. PMID 16773644
- [Background] Peterson DS, Fling BW, Mancini M, Cohen RG, Nutt JG, Horak FB. Dual-task interference and brain structural connectivity in people with Parkinson's disease who freeze. J Neurol Neurosurg Psychiatry. 2015 Jul;86(7):786-92. doi: 10.1136/jnnp-2014-308840. Epub 2014 Sep 15. PMID 25224677
- [Background] Plotnik M, Giladi N, Hausdorff JM. Is freezing of gait in Parkinson's disease a result of multiple gait impairments? Implications for treatment. Parkinsons Dis. 2012;2012:459321. doi: 10.1155/2012/459321. Epub 2012 Jan 12. PMID 22288021
- [Background] Nonnekes J, Janssen AM, Mensink SH, Oude Nijhuis LB, Bloem BR, Snijders AH. Short rapid steps to provoke freezing of gait in Parkinson's disease. J Neurol. 2014 Sep;261(9):1763-7. doi: 10.1007/s00415-014-7422-8. Epub 2014 Jun 24. PMID 24957299
- [Background] Morris M, Iansek R, Matyas T, Summers J. Abnormalities in the stride length-cadence relation in parkinsonian gait. Mov Disord. 1998 Jan;13(1):61-9. doi: 10.1002/mds.870130115. PMID 9452328
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Peto V, Jenkinson C, Fitzpatrick R, Greenhall R. The development and validation of a short measure of functioning and well being for individuals with Parkinson's disease. Qual Life Res. 1995 Jun;4(3):241-8. doi: 10.1007/BF02260863. PMID 7613534